CLINICAL TRIAL: NCT02939352
Title: The Effects of a Single Session of Real Versus Sham Theta Burst Stimulation on the Brain Response to Drug-cues
Brief Title: The Effects of Theta Burst Stimulation on the Brain Response to Drug and Alcohol Cues
Acronym: addictionTBS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 30506
Record Dates: First submitted 2015-09-28; First posted 2016-10-20 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Alcoholism; Cocaine Addiction; Drug Addiction
Keywords: Transcranial Magnetic Stimulation; Magnetic Resonance Imaging; MRI, Functional
MeSH Terms: conditions — Alcoholism; Cocaine-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cocaine Users (Experimental): Participants will receive Real continuous Theta Burst Stimulation to the left frontal pole/medial prefrontal cortex. Participants will also receive Sham continuous Theta Burst Stimulation to the left frontal pole/medial prefrontal cortex.
  Interventions: Device: Real continuous Theta Burst Stimulation; Device: Sham continuous Theta Burst Stimulation
- Alcohol Users (Experimental): Participants will receive Real continuous Theta Burst Stimulation to the left frontal pole/medial prefrontal cortex. Participants will also receive Sham continuous Theta Burst Stimulation to the left frontal pole/medial prefrontal cortex.
  Interventions: Device: Real continuous Theta Burst Stimulation; Device: Sham continuous Theta Burst Stimulation

INTERVENTIONS:
Device: Real continuous Theta Burst Stimulation — Continuous Theta Burst stimulation delivered
Device: Sham continuous Theta Burst Stimulation — active sham Continuous Theta Burst stimulation delivered

SUMMARY:
High relapse rates among substance dependent individuals are likely due to a combination of factors that involve limbic circuits in the brain involved in craving, including vulnerability to salient cues. Emerging data suggests that non-invasive, targeted brain stimulation may be able to modulate activity in these circuits and decrease craving. The primary goal of this pilot study is to determine the extent to which a single session of continuous theta burst stimulation to the medial prefrontal cortex can attenuate limbic circuitry involved in craving among cocaine users and alcohol users. This will be tested through a double-blind,sham-controlled brain stimulation and brain imaging study in a cohort of polysubstance abusers and alcohol users.

DETAILED DESCRIPTION:
This parent protocol contains two components - one of which is targeting cocaine users, the other of which is targeting heavy alcohol users (who will also serve as an appropriate control group for the cocaine users - who typically have comorbid alcohol use disorders). All participants will receive one session of real and one session of sham (randomized) continuous theta burst stimulation (TBS).TBS is a form of non-invasive transcranial magnetic stimulation (TMS).Continuous TBS is designed to lower cortical excitability, and requires a shorter stimulation period than typical low frequency TMS. The investigators will test the hypotheses that stimulation over the medial prefrontal cortex will attenuate activity in the medial prefrontal cortex (Aim 1), using single pulse TMS in the magnetic resonance imaging scanner. Through this innovative technique it is possible to apply a single pulse of TMS to the medial prefrontal cortex and model the hemodynamic response at the stimulation site as well as monosynaptic target regions, including the striatum. The investigators will also investigate the effect of TBS on neural response to drug cues (Aim 2). The results of these aims will be further correlated with self-reported assessments of craving throughout each experimental visit. These data will be preliminary data for a subsequent R01 focused on the sustained effects of multiple sessions of TBS and their efficacy in lowering craving for extended periods of time in treatment-seekers.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-55
* Non-treatment seeking cocaine users (with or without comorbid alcohol use disorder)
* Current alcohol use greater than 20 standard drinks per week
* Current DSM-V Alcohol Use Disorder diagnosis, including the loss of control item
* Currently not engaged in, and do not want treatment for, alcohol related problems
* Able to read and understand questionnaires and informed consent
* Lives within 50 miles of the study site

Exclusion Criteria [These are listed in greater detail in the CIA Core]:

* Any current DSM-V Axis I diagnosis except Alcohol, Cocaine, or Nicotine Use Disorder
* Current or past substance dependence criteria other than cocaine, marijuana, or alcohol, smoking >1 pack of cigarettes per day
* Current use of any psychoactive substance except cocaine, nicotine, and marijuana or medications as evidenced by self-report or urine drug screen
* Current breath alcohol concentration >0.002
* Positive urine drug screen for stimulants (including cocaine, amphetamine, methamphetamine, etc.) at the Scanning/Stimulation visits and signs of alcohol withdrawal. Based on the sensitivity of this test, this will require that the participants abstain from cocaine use for 48 hours prior to the intervention
* History of seizures or migraine headaches
* History of head trauma or epilepsy
* Violation of other magnetic resonance imaging safety measures
* Current suicidal or homicidal ideation
* Presence of ferrous metal in the body, as evidenced by metal screening and self-report
* Severe claustrophobia or extreme obesity that preclude placement in the MRI scanner
* For female participants, pregnancy, as evidenced by a urine pregnancy test administered on the day of the scanning session

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percent Blood Oxygen-Level Dependent (BOLD) signal change in the Medial Prefrontal Cortex (MPFC) | 1 hour

SECONDARY OUTCOMES:
Self reported craving | 1 hour
  Tiffany Craving Scale
Percent Blood Oxygen-Level Dependent (BOLD) signal change in the Striatum | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A Hanlon, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kearney-Ramos TE, Dowdle LT, Lench DH, Mithoefer OJ, Devries WH, George MS, Anton RF, Hanlon CA. Transdiagnostic Effects of Ventromedial Prefrontal Cortex Transcranial Magnetic Stimulation on Cue Reactivity. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jul;3(7):599-609. doi: 10.1016/j.bpsc.2018.03.016. Epub 2018 Apr 10. PMID 29776789